CLINICAL TRIAL: NCT01062698
Title: The Contribution of Intra-arterial Thrombectomy in Acute Ischemic Stroke in Patients Treated With Intravenous Thrombolysis
Brief Title: Trial and Cost Effectiveness Evaluation of Intra-arterial Thrombectomy in Acute Ischemic Stroke
Acronym: THRACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Efficacy
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Directeur de la Recherche et de l'Innovation, Professor Serge BRACARD, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-A00753-54
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cerebral Stroke; Cerebrovascular Accident
Keywords: mechanical Thrombectomy; CVA (Cerebrovascular Accident); Cerebrovascular Accident, Acute
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Solitaire composite resin

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- IV thrombolysis + thrombectomy (Active Comparator)
  Interventions: Drug: Alteplase (rt-PA)/Actilyse; Procedure: Mechanic thrombectomy (MERCI, PENUMBRA, CATCH, SOLITAIRE)
- IV thrombolysis (Active Comparator)
  Interventions: Drug: Alteplase (rt-PA)/Actilyse

INTERVENTIONS:
Drug: Alteplase (rt-PA)/Actilyse — Injection of 0.9 mg/kg for 60min with an initial 10% bolus injection.
Procedure: Mechanic thrombectomy (MERCI, PENUMBRA, CATCH, SOLITAIRE) — Mechanic thrombectomy
  Arms: IV thrombolysis + thrombectomy

SUMMARY:
THRACE is a controled, multicenter and randomized trial.

The primary objective of this study is to determine whether a combined approach intravenous thrombolysis (IV) + Mechanical thrombectomy is superior to the reference treatment with IV thrombolysis alone, in the 3 hours of onset of symptoms in patients with occlusion of proximal cerebral arteries and with a neurological impairment accident (National Institutes of Health Stroke Scale [NIHSS] ≥ 10).

The second objective is to determine the cost-effectiveness of this procedure compared to the standard (IV thrombolysis). The assumption is that the combined approach, by improving the clinical outcome and speed recovery, allows for lower overall costs to the IV thrombolysis in 3 months and less than or at worst neutral to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 10<=NIHSS Score=<25
* Symptoms onset less than 4 hours
* Occlusion of the intracranial carotid, the middle cerebral artery (M1) or the upper third of the basilar

Exclusion Criteria:

* Contraindications for intravenous thrombolysis
* Occlusion or stenosis of the pre-occlusive cervical internal carotid artery ipsilateral to the lesion
* Any cause local prohibiting femoral catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12; Study Completion 2016-03

PRIMARY OUTCOMES:
Modified Rankin Score (mRs ) | 3 months after treatment

SECONDARY OUTCOMES:
Quality of Life (Euroqol EQ-5D) | 3 months after treatment
Barthel Score | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Serge Bracard, Pr, Principal Investigator — Central Hospital Nancy France (HNF)
Locations (1):
- Central Hospital Nancy (Central HNF), Nancy, France

REFERENCES:
- [Derived] Agbonon R, Forestier G, Bricout N, Benhassen W, Turc G, Bretzner M, Pasi M, Benzakoun J, Seners P, Derraz I, Legrand L, Trystram D, Rodriguez-Regent C, Charidimou A, Rost NS, Bracard S, Cordonnier C, Eker OF, Oppenheim C, Naggara O, Henon H, Boulouis G. Cerebral microbleeds and risk of symptomatic hemorrhagic transformation following mechanical thrombectomy for large vessel ischemic stroke. J Neurol. 2024 May;271(5):2631-2638. doi: 10.1007/s00415-024-12205-7. Epub 2024 Feb 14. PMID 38355868
- [Derived] Janvier P, Kerleroux B, Turc G, Pasi M, Farhat W, Bricout N, Benzakoun J, Legrand L, Clarencon F, Bracard S, Oppenheim C, Boulouis G, Henon H, Naggara O, Ben Hassen W. TAGE Score for Symptomatic Intracranial Hemorrhage Prediction After Successful Endovascular Treatment in Acute Ischemic Stroke. Stroke. 2022 Sep;53(9):2809-2817. doi: 10.1161/STROKEAHA.121.038088. Epub 2022 Jun 14. PMID 35698971
- [Derived] Riou-Comte N, Gory B, Soudant M, Zhu F, Xie Y, Humbertjean L, Mione G, Oppenheim C, Guillemin F, Bracard S, Richard S; THRACE investigators. Clinical imaging factors of excellent outcome after thrombolysis in large-vessel stroke: a THRACE subgroup analysis. Stroke Vasc Neurol. 2021 Dec;6(4):631-639. doi: 10.1136/svn-2020-000852. Epub 2021 Jun 8. PMID 34103393
- [Derived] Derraz I, Pou M, Labreuche J, Legrand L, Soize S, Tisserand M, Rosso C, Piotin M, Boulouis G, Oppenheim C, Naggara O, Bracard S, Clarencon F, Lapergue B, Bourcier R; ASTER and the THRACE Trials Investigators. Clot Burden Score and Collateral Status and Their Impact on Functional Outcome in Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2021 Jan;42(1):42-48. doi: 10.3174/ajnr.A6865. Epub 2020 Nov 12. PMID 33184069
- [Derived] Boulouis G, Bricout N, Benhassen W, Ferrigno M, Turc G, Bretzner M, Benzakoun J, Seners P, Personnic T, Legrand L, Trystram D, Rodriguez-Regent C, Charidimou A, Rost NS, Bracard S, Cordonnier C, Oppenheim C, Naggara O, Henon H. White matter hyperintensity burden in patients with ischemic stroke treated with thrombectomy. Neurology. 2019 Oct 15;93(16):e1498-e1506. doi: 10.1212/WNL.0000000000008317. Epub 2019 Sep 13. PMID 31519778
- [Derived] Provost C, Soudant M, Legrand L, Ben Hassen W, Xie Y, Soize S, Bourcier R, Benzakoun J, Edjlali M, Boulouis G, Raoult H, Guillemin F, Naggara O, Bracard S, Oppenheim C. Magnetic Resonance Imaging or Computed Tomography Before Treatment in Acute Ischemic Stroke. Stroke. 2019 Mar;50(3):659-664. doi: 10.1161/STROKEAHA.118.023882. PMID 30744542
- [Derived] Achit H, Soudant M, Hosseini K, Bannay A, Epstein J, Bracard S, Guillemin F; THRACE Investigators. Cost-Effectiveness of Thrombectomy in Patients With Acute Ischemic Stroke: The THRACE Randomized Controlled Trial. Stroke. 2017 Oct;48(10):2843-2847. doi: 10.1161/STROKEAHA.117.017856. Epub 2017 Sep 15. PMID 28916667
- [Derived] Bracard S, Ducrocq X, Mas JL, Soudant M, Oppenheim C, Moulin T, Guillemin F; THRACE investigators. Mechanical thrombectomy after intravenous alteplase versus alteplase alone after stroke (THRACE): a randomised controlled trial. Lancet Neurol. 2016 Oct;15(11):1138-47. doi: 10.1016/S1474-4422(16)30177-6. Epub 2016 Aug 23. PMID 27567239